CLINICAL TRIAL: NCT04613089
Title: Natural History and Long Term Clinical Assessments of All Forms of Neuronal Ceroid Lipofuscinoses - Capturing Key Symptoms and Disease Progression as Part of the Independent, International NCL DEM-CHILD Patient Database
Brief Title: Natural History and Longitudinal Clinical Assessments in NCL / Batten Disease, the International DEM-CHILD Database
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Angela Schulz, MD, PhD, Head of NCL Specialty Clinic, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: DEM-CHILD2020
Record Dates: First submitted 2020-09-10; First posted 2020-11-03 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Neuronal Ceroid Lipofuscinosis; Batten Disease; CLN1 Disease; CLN2 Disease; CLN3 Disease; CLN4 Disease; CLN5 Disease; CLN6 Disease; CLN7 Disease; CLN8 Disease; CLN10 Disease; CLN11 Disease; CLN12 Disease; CLN13 Disease; CLN14 Disease
Keywords: INCL; LINCL; VLINCL; JNCL; ANCL; NCL; CLN; Batten; Childhood Dementia; Lysosomal Storage Diseases; Neurodegenerative Diseases; Neurodegenerative Disorders; Metabolic Disorders; PME; EPMR; SCAR7; SGSH; PPT1; Haltia-Santavuori Disease; TPP1; Jansky-Bielschowsky Disease; Spielmeyer-Vogt-Sjögren-Batten Disease; DNAJC5; Parry Disease; Kufs Disease Type A; MFSD8; CTSD; GRN; ATP13A2; Kufor-Rakeb Syndrome; CTSF; Kufs Disease Type B; KCTD7
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses; Ceroid lipofuscinosis, neuronal 5; Lysosomal Storage Diseases; Neurodegenerative Diseases; Metabolic Diseases; Kufor-Rakeb syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — All available Biomaterials from diagnostic approach and routine clinical care are collected (e.g. blood, urine, skin cells, CSF, other..).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- CLN1 Disease, Haltia-Santavuori Disease: Patients with genetic mutations in the CLN1/PPT1 gene, causing a lysosomal enzyme deficiency of PPT1.
  Interventions: Other: Natural History
- CLN2 Disease, Jansky-Bielschowsky Disease: Patients with genetic mutations in the CLN2/TPP1 gene, causing a lysosomal enzyme deficiency of TTP1.
  Interventions: Other: Natural History
- CLN2 Disease - ERT (Brineura) treated: Patients with genetic mutations in the CLN2/TPP1 gene, causing a lysosomal enzyme deficiency of TTP1, previously and/or currently receiving enzyme-replacement therapy (ERT) with Cerliponase alpha (Brineura).
  Interventions: Other: Natural History
- CLN3 Disease, Spielmeyer-Vogt-Sjögren-Batten Disease: Patients with genetic mutations in the CLN3 gene.
  Interventions: Other: Natural History
- CLN4 disease, Parry disease: Patients with genetic mutations in the CLN4/DNAJC5 gene.
  Interventions: Other: Natural History
- CLN5 Disease: Patients with genetic mutations in the CLN5 gene.
  Interventions: Other: Natural History
- CLN6 Disease, Kufs Disease Type A: Patients with genetic mutations in the CLN6 gene.
  Interventions: Other: Natural History
- CLN7 Disease: Patients with genetic mutations in the CLN7/MFSD8 gene.
  Interventions: Other: Natural History
- CLN8 Disease: Patients with genetic mutations in the CLN8 gene.
  Interventions: Other: Natural History
- CLN10 Disease: Patients with genetic mutations in the CLN10/CTSD gene, causing a lysosomal enzyme deficiency of Cathepsin D.
  Interventions: Other: Natural History
- CLN11 Disease: Patients with genetic mutations in the CLN11/GRN gene.
  Interventions: Other: Natural History
- CLN12 Disease: Patients with genetic mutations in the CLN12/ATP13A2 gene.
  Interventions: Other: Natural History
- CLN13 Disease, Kufs Disease Type B: Patients with genetic mutations in the CLN13/CTSF gene, causing a lysosomal enzyme deficiency of Cathepsin F.
  Interventions: Other: Natural History
- CLN14 Disease: Patients with genetic mutations in the CLN14/KCTD7 gene.
  Interventions: Other: Natural History

INTERVENTIONS:
Other: Natural History — Natural History and Clinical Follow Up.

SUMMARY:
This is an observational study that aims at assessing the natural history of NCL diseases as part of the international DEM-CHILD Database.

1. Patient data are collected from medical records, patient questionnaires and routine follow up clinical examinations with focus on assessing progression in key areas of disease such as motor, language, cognition, seizures, vision, and behavior.
2. A local biorepository of samples from genetically defined NCL patients will be established as well as a virtual biorepository within the DEM-CHILD DB to be able to easily localize international availability of patient samples.

DETAILED DESCRIPTION:
NCLs (Neuronal Ceroid Lipofuscinoses) are a group of rare, inherited, neurodegenerative disorders, also known as Batten disease. Until now, 13 different genes causing different subtypes of disease are known. The genetic mutations cause a symptom complex of progressive loss of acquired skills in the domains of motor function, cognition and visual function, leading to ataxia, movement disorder, dementia, blindness and seizures. In the area of genetic testing, variable clinical phenotypes become more and more prevalent. The disease-mechanisms as well as the exact clinical course of the diseases are currently still not fully understood and documented. Although descriptions of the clinical spectrums exist, the natural history needs to be defined as accurately as possible. These data are urgently needed as clinical control data helping to test the therapeutic efficacy of emerging experimental therapies.

Since samples of genetically defined patients are rare and therefore limited for research, there is an urgent need for researchers to localize and access samples internationally. With the establishment of a local NCL-biorepository and virtual sample localization internationally, scientists worldwide may have a faster way to access needed samples for advancing research.

Any NCL patient with a confirmed molecular diagnosis can join the retrospective and prospective natural history data collection. It is also possible for families with already deceased patients to participate in the retrospective analysis part of the data collection if the genetic mutation is known.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a confirmed molecular diagnosis of a form of NCL Disease

Additional inclusion criteria for Group/Cohort: "CLN2 Disease - ERT (Brineura) Treated":

* Documented diagnosis of TPP1 deficiency
* Previous or current treatment with intracerebroventricular ERT with cerliponase alpha
* Patients that are currently participating in post-marketing studies will be allowed to participate.

Exclusion Criteria:

- Patients with no confirmed molecular diagnosis of a form of NCL Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, Adolescents, Adults
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2050-04-08 (Estimated); Study Completion 2050-04-08 (Estimated)

PRIMARY OUTCOMES:
Identification of key symptoms of disease, natural history of disease progression and development of quantitative tools for rating disease progression that can be used as therapeutic outcome measures for emerging experimental therapies. | Up to 30 years
  Evaluation of Medical history from patient interviews and medical chart review. Evaluating data from clinical routine follow up exams (e.g. brain imaging MRI, ophthalmologic assessments, OCT, EEG, cardiology assessments, cognitive assessments, developmental scales, clinical rating scales).
Establish well characterized Natural History Cohorts from genetically defined NCL patients to provide these as Natural History Control Cohorts for new experimental therapy trials. | Up to 30 years
  Analysis of retrospective and prospective data from patient interviews and medical chart review as well as clinical routine follow up exams (e.g. brain imaging MRI, ophthalmologic assessments, OCT, EEG, cardiology assessments, cognitive assessments, developmental scales, clinical rating scales).

SECONDARY OUTCOMES:
Establish a biorepository of samples from genetically defined NCL patients. | Up to 30 years
  - Collection of biospecimens that have been collected within treatment as part of standard of care.
Establish a virtual biorepository from genetically defined NCL patients within the DEM-CHILD Database. | Up to 30 years
  Datacollection of available biospecimens from genetically defined NCL patients and the collecting center contacts within the DEM-CHILD DB.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Schulz, MD, PhD, Principal Investigator — Head of NCL-Specialty Clinic
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
The goal of the independent international DEM-CHILD DB is to collect high quality natural history data of NCL patients. The independent nature of the database allows to make data available for international research on treatment evaluation and development.
Supporting Information: Study Protocol, ICF
Access Criteria: Upon written formal request. Project description of anticipated data usage needed. Specifications for exact data access (type of NCL, retrospective or prospective data, data items) and data transfer (one-time transfer, longitudinal access) must be declared. Data transfer agreements detailing the above will need to be in place with the respective data-entering center who has full data ownership.

REFERENCES:
- [Background] Rietdorf K, Coode EE, Schulz A, Wibbeler E, Bootman MD, Ostergaard JR. Cardiac pathology in neuronal ceroid lipofuscinoses (NCL): More than a mere co-morbidity. Biochim Biophys Acta Mol Basis Dis. 2020 Sep 1;1866(9):165643. doi: 10.1016/j.bbadis.2019.165643. Epub 2019 Dec 19. PMID 31863828
- [Background] Nickel M, Simonati A, Jacoby D, Lezius S, Kilian D, Van de Graaf B, Pagovich OE, Kosofsky B, Yohay K, Downs M, Slasor P, Ajayi T, Crystal RG, Kohlschutter A, Sondhi D, Schulz A. Disease characteristics and progression in patients with late-infantile neuronal ceroid lipofuscinosis type 2 (CLN2) disease: an observational cohort study. Lancet Child Adolesc Health. 2018 Aug;2(8):582-590. doi: 10.1016/S2352-4642(18)30179-2. Epub 2018 Jul 2. PMID 30119717
- [Background] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815
- [Background] Gardner E, Bailey M, Schulz A, Aristorena M, Miller N, Mole SE. Mutation update: Review of TPP1 gene variants associated with neuronal ceroid lipofuscinosis CLN2 disease. Hum Mutat. 2019 Nov;40(11):1924-1938. doi: 10.1002/humu.23860. Epub 2019 Jul 26. PMID 31283065
- [Background] Fietz M, AlSayed M, Burke D, Cohen-Pfeffer J, Cooper JD, Dvorakova L, Giugliani R, Izzo E, Jahnova H, Lukacs Z, Mole SE, Noher de Halac I, Pearce DA, Poupetova H, Schulz A, Specchio N, Xin W, Miller N. Diagnosis of neuronal ceroid lipofuscinosis type 2 (CLN2 disease): Expert recommendations for early detection and laboratory diagnosis. Mol Genet Metab. 2016 Sep;119(1-2):160-7. doi: 10.1016/j.ymgme.2016.07.011. Epub 2016 Jul 25. PMID 27553878
- [Background] Simonati A, Williams RE, Nardocci N, Laine M, Battini R, Schulz A, Garavaglia B, Moro F, Pezzini F, Santorelli FM. Phenotype and natural history of variant late infantile ceroid-lipofuscinosis 5. Dev Med Child Neurol. 2017 Aug;59(8):815-821. doi: 10.1111/dmcn.13473. Epub 2017 May 25. PMID 28542837
- [Background] Lebrun AH, Storch S, Ruschendorf F, Schmiedt ML, Kyttala A, Mole SE, Kitzmuller C, Saar K, Mewasingh LD, Boda V, Kohlschutter A, Ullrich K, Braulke T, Schulz A. Retention of lysosomal protein CLN5 in the endoplasmic reticulum causes neuronal ceroid lipofuscinosis in Asian sibship. Hum Mutat. 2009 May;30(5):E651-61. doi: 10.1002/humu.21010. PMID 19309691
- [Background] Williams RE, Adams HR, Blohm M, Cohen-Pfeffer JL, de Los Reyes E, Denecke J, Drago K, Fairhurst C, Frazier M, Guelbert N, Kiss S, Kofler A, Lawson JA, Lehwald L, Leung MA, Mikhaylova S, Mink JW, Nickel M, Shediac R, Sims K, Specchio N, Topcu M, von Lobbecke I, West A, Zernikow B, Schulz A. Management Strategies for CLN2 Disease. Pediatr Neurol. 2017 Apr;69:102-112. doi: 10.1016/j.pediatrneurol.2017.01.034. Epub 2017 Feb 4. PMID 28335910
- [Background] Kohlschutter A, Schulz A, Bartsch U, Storch S. Current and Emerging Treatment Strategies for Neuronal Ceroid Lipofuscinoses. CNS Drugs. 2019 Apr;33(4):315-325. doi: 10.1007/s40263-019-00620-8. PMID 30877620
- [Background] Lobel U, Sedlacik J, Nickel M, Lezius S, Fiehler J, Nestrasil I, Kohlschutter A, Schulz A. Volumetric Description of Brain Atrophy in Neuronal Ceroid Lipofuscinosis 2: Supratentorial Gray Matter Shows Uniform Disease Progression. AJNR Am J Neuroradiol. 2016 Oct;37(10):1938-1943. doi: 10.3174/ajnr.A4816. Epub 2016 May 26. PMID 27231226
- [Background] Dulz S, Wagenfeld L, Nickel M, Richard G, Schwartz R, Bartsch U, Kohlschutter A, Schulz A. Novel morphological macular findings in juvenile CLN3 disease. Br J Ophthalmol. 2016 Jun;100(6):824-8. doi: 10.1136/bjophthalmol-2015-307320. Epub 2015 Oct 20. PMID 26486417
- [Background] Dulz S, Atiskova Y, Wibbeler E, Wildner J, Wagenfeld L, Schwering C, Nickel M, Bartsch U, Spitzer MS, Schulz A. An Ophthalmic Rating Scale to Assess Ocular Involvement in Juvenile CLN3 Disease. Am J Ophthalmol. 2020 Dec;220:64-71. doi: 10.1016/j.ajo.2020.07.015. Epub 2020 Jul 21. PMID 32707205
- [Background] Mole SE, Anderson G, Band HA, Berkovic SF, Cooper JD, Kleine Holthaus SM, McKay TR, Medina DL, Rahim AA, Schulz A, Smith AJ. Clinical challenges and future therapeutic approaches for neuronal ceroid lipofuscinosis. Lancet Neurol. 2019 Jan;18(1):107-116. doi: 10.1016/S1474-4422(18)30368-5. Epub 2018 Nov 21. PMID 30470609
- [Background] Bergholz R, Kohlschutter A, Schulz A, Hubert W, Ruther K. Phenotyping heterozygous carriers of juvenile neuronal ceroid lipofuscinosis with CLN3 mutations. Graefes Arch Clin Exp Ophthalmol. 2015 Aug;253(8):1245-50. doi: 10.1007/s00417-014-2814-0. Epub 2014 Oct 22. PMID 25338278
- [Background] Schulz A, Kohlschutter A, Mink J, Simonati A, Williams R. NCL diseases - clinical perspectives. Biochim Biophys Acta. 2013 Nov;1832(11):1801-6. doi: 10.1016/j.bbadis.2013.04.008. Epub 2013 Apr 17. PMID 23602993
- [Background] Paniagua Bravo A, Forkert ND, Schulz A, Lobel U, Fiehler J, Ding X, Sedlacik J, Rosenkranz M, Goebell E. Quantitative t2 measurements in juvenile and late infantile neuronal ceroid lipofuscinosis. Clin Neuroradiol. 2013 Sep;23(3):189-96. doi: 10.1007/s00062-012-0189-3. Epub 2012 Dec 23. PMID 23263384
- [Background] Kousi M, Anttila V, Schulz A, Calafato S, Jakkula E, Riesch E, Myllykangas L, Kalimo H, Topcu M, Gokben S, Alehan F, Lemke JR, Alber M, Palotie A, Kopra O, Lehesjoki AE. Novel mutations consolidate KCTD7 as a progressive myoclonus epilepsy gene. J Med Genet. 2012 Jun;49(6):391-9. doi: 10.1136/jmedgenet-2012-100859. PMID 22693283
- [Derived] Dulz S, Schwering C, Wildner J, Spartalis C, Schuettauf F, Bartsch U, Wibbeler E, Nickel M, Spitzer MS, Atiskova Y, Schulz A. Ongoing retinal degeneration despite intraventricular enzyme replacement therapy with cerliponase alfa in late-infantile neuronal ceroid lipofuscinosis type 2 (CLN2 disease). Br J Ophthalmol. 2023 Oct;107(10):1478-1483. doi: 10.1136/bjo-2022-321260. Epub 2022 Jun 30. PMID 35772852